CLINICAL TRIAL: NCT02911025
Title: Effects of Clobazam on Sleep and Daytime Function in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Pavlova, Milena,M.D., Assistant Professor, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2014P001657
Record Dates: First submitted 2016-01-11; First posted 2016-09-22 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy
Keywords: epilepsy; sleep; antiepileptic drugs
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Treated With Clobazam: Single group, patients treated with clobazam by their treating physician (no interventions from PI), followed longitudinally for 1 week after reaching effective clobazam dose.

SUMMARY:
The purpose of this study is to monitor the effect of Clobazam on sleep and daytime alertness in people with Epilepsy.

DETAILED DESCRIPTION:
Many studies show that patients with epilepsy frequently have disrupted sleep, as well as a high level of daytime sleepiness. This may be due to a sleep disorder, nighttime seizures that lead to disrupted sleep, and other abnormalities. Sleep complaints are widely reported among patients with various epilepsy syndromes.

Anti-seizure treatments may affect sleep. Effects vary by type of medication and other health issues. Generally, with improvement of seizure control, the sleep cycle improves and becomes more regular. However, some anti-seizure medications have been associated with insomnia. There have been studies that looked at sleep in relation to some anti-seizure medications. However, there are no currently available published reports on the effect of Clobazam (Onfi) on sleep.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or older
* diagnosis of epilepsy who are being considered for treatment with Clobazam

Exclusion Criteria:

* known untreated moderate or severe sleep apnea
* major circadian rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Epilepsy who have recently been started on Clobazam (Onfi)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milena Pavlova, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Jamaica Plain, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Treated With Clobazam
Started | 13
Completed | 10
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With Clobazam
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep (Total Sleep Time) in Patients With Epilepsy Treated With Clobazam
Description: The change in total sleep time in patients with epilepsy treat with clobazam one week after reaching effective clobazam dose
Time Frame: 1 week after reaching effective clobazam dose
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients Treated With Clobazam
Number analyzed (Participants) | 13
minutes
  Baseline Phase | 493.2 (457.9)
  Treatment Phase | 457.9 (23.9)

2. Secondary Outcome: Change in Sleep (Wake After Sleep Onset) in Patients With Epilepsy Treated With Clobazam
Description: The change in wake after sleep onset (WASO) in patients with epilepsy treat with clobazam one week after reaching effective clobazam dose
Time Frame: 1 week after reaching effective clobazam dose
Measure: Mean (Standard Deviation); unit: count of awakenings
Arm/Group | Patients Treated With Clobazam
Number analyzed (Participants) | 13
count of awakenings
  Baseline Phase | 50.2 (6.9)
  Treatment Phase | 37.3 (3.5)

ADVERSE EVENTS:
Time Frame: Each patient was followed for one week during the treatment phase.
Arm/Group | Patients Treated With Clobazam
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Clobazam (N=13)
Sedation Side Effect (Product Issues) | 1 (1) — Patient felt sedation when taking this medication and did not enjoy it.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02911025/Prot_SAP_000.pdf